CLINICAL TRIAL: NCT05810402
Title: Liver Cancer and Immunotherapy : Clinical Relevance of LIquid BioPSY
Brief Title: Liver Cancer and Immunotherapy in the Liquid Biopsy Era
Acronym: LILIPSY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL22_0514
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Hepatocellular Carcinoma; BCLC Stage B Hepatocellular Carcinoma; BCLC Stage C Hepatocellular Carcinoma; Immune Checkpoint Inhibitor; Liquid Biopsy
Keywords: Hepatocellular Carcinoma; BCLC Stage B and C; Immune Checkpoint Inhibitor; Liquid Biopsy; Precision Medicine
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Liquid Biopsy; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Homogenous cohort of BCLC Stage B and C hepatocellular carcinoma patients that will undergo immunotherapy +/- anti-angiogenic agent (bevacizumab)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BCLC B and C HCC patients (Experimental): For each participant, 30mL of blood will be collected at inclusion/before treatment initiation (baseline) and during standard of care follow-up.
  The blood sample will be taken, in consultation or in outpatient clinic during a blood test for health purposes.
  Interventions: Biological: Liquid Biopsy

INTERVENTIONS:
Biological: Liquid Biopsy — 30mL blood sample:
  * 1 x 10mL CellSave tube specifically designed for the collection and preservation of CTCs for CellSearch® analysis
  * 1 EDTA tube for PBMCs isolation and circulating immune cells study (5mL),
  * 2 EDTA tubes and 1 dry tube (15mL) for the preparation of the biobank (serum, plasma and cell).
  Other Names: Blood sample

SUMMARY:
The goal of this prospective clinical trial is to identify a predictive biomarker in patients with advanced HCC (stage B and C) using a combinatorial approach of the liquid biopsy.

The main questions it aims to answer are:

* Is multi-omic liquid biopsy approach able to identify a strong predictive biomarker of immunotherapy efficiency?
* Is there a correlation between tissue biopsy (PD-L1 tissue level of expression) and liquid biopsy (detection of CTC expressing PD-L1) in HCC patients?

Participants blood will be collected at several time points.

DETAILED DESCRIPTION:
In solid cancers, some more aggressive tumor cells actively detach from the primary lesion and then travel through the circulating compartment to reach distant organs and form micro-metastases. Detecting CTCs in the blood is also relevant for assessing tumor progression, prognosis and therapeutic follow-up. The non-invasive, highly sensitive for CTCs analysis is called "liquid biopsy". Over the past few years, a multi-analyses approach (CTCs, circulating tumor DNA, extracellular vesicles, miRNA...) of liquid biopsy has been developed.

Hepatocellular carcinoma (HCC) is the predominant pathological type of primary liver cancer. It represents the sixth most common incidence worldwide and the third most common cause of cancer mortality.

Since 2021, the gold standard treatment for patients with advanced and/or unresectable HCC is the combination of atezolizumab (anti-PD-L1) and bevacizumab (VEGF inhibitor) in cases where chemoembolization is not indicated (patients with lymph node invasion and/or distant lesions or patients with portal flow abnormality). Indeed, this therapy offers a significant benefit in overall survival (19.2 vs 13.4 months, HR 0.66, p<0.0009) as well as in progression-free survival (6.9 vs 4.3 months, HR 0.65, p=0.0001). However, to date, there is no predictive biomarker for the efficacy of immune checkpoint inhibitors (ICI)

The purpose of this research project is to identify a predictive biomarker in patients with advanced HCC (stage B and C) using a combinatorial approach of the liquid biopsy (CTC, CTC expressing PD-L1, immune cell profiling).

ELIGIBILITY:
Inclusion Criteria:

* Patients of at least 18 years old,
* Patients with advanced hepatocellular carcinoma or HCC with indication for first-line PD-1 or PD-L1 immunotherapy in MDT, without prior systemic therapy,
* The diagnosis of HCC is established according to imaging criteria (LI-RADSv2018 criteria) or after histological evidence,
* Advanced HCC defined by BCLC stages B and C,
* Patients with oral consent.

Exclusion Criteria:

* Administration of a previous systemic anti-tumor treatment (immunotherapy or chemotherapy or targeted therapy)
* No personal history of neoplasia in the previous 5 years
* No personal history of systemic inflammatory diseases
* No immunosuppressive treatment or treatment that could modify immunity (anti-TNF...)
* No affiliation or non-beneficiary of a Social Security system;
* Vulnerable persons according to article L1121-6 of the CSP ;
* Persons of full age who are protected or unable to give their consent according to article L1121-8 of the CSP;
* Pregnant or breastfeeding women according to article L1121-5 of the CSP.
* Non-inclusion due to follow-up difficulties (transfer, insufficient motivation, poor compliance, priority associated pathology in care, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with CTCs-PD-L1+ by CellSearch® technique | At inclusion
  A CTC is being defined as: EpCAM(+)/PanCK(+)/Dapi(+)/CD45(-). The PD-L1 status will be observed only on these cells. CTC-PD-L1- = 0 vs CTC-PD-L1+ ≥1

SECONDARY OUTCOMES:
Number of CTCs-PD-L1+ measured by CellSearch® technique | At inclusion
  0 vs. 1 vs. 2-3 vs. 4 vs. ≥5
Presence of CTCs at inclusion by CellSearch® technique | At inclusion
  Percentage of patients with CTCs
Number of CTCs measured by CellSearch® technique | At inclusion
  0 vs 1 vs 2-3 vs 4 vs ≥5
Immune profiling | 24 month follow up
  FACS study of immune system cells (T cells, NK cells, B cells, macrophages, immune-checkpoint and platelets)
Expression of PD-L1 by immuno-histochemical analysis of tissue samples | At inclusion
  PD-L1 expression on biopsy or surgical specimen previously preserved in the Montpellier University Hospital tumor library
Tumor control defined by mRECIST criteria | 24 month follow up
  Best response: complete response + partial response + stable vs progression
Tumor control defined by RECIST criteria | 24 month follow up
  Best response: complete response + partial response + stable vs progression
Overall Survival | 24 month follow-up
  Time from immunotherapy start date to date of death from any cause
Progression Free Survival | 24 month follow-up
  Time from immunotherapy start date to date of first progression or date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Alix-Panabières, Ph.D., Study Director — University Hospital, Montpellier; Thomas Bardol, M.D., Principal Investigator — University Hospital, Montpellier
Locations (1):
- CHU Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pantel K, Alix-Panabieres C. Tumour microenvironment: informing on minimal residual disease in solid tumours. Nat Rev Clin Oncol. 2017 Jun;14(6):325-326. doi: 10.1038/nrclinonc.2017.53. Epub 2017 Apr 11. No abstract available. PMID 28397823
- [Background] Meng S, Tripathy D, Frenkel EP, Shete S, Naftalis EZ, Huth JF, Beitsch PD, Leitch M, Hoover S, Euhus D, Haley B, Morrison L, Fleming TP, Herlyn D, Terstappen LW, Fehm T, Tucker TF, Lane N, Wang J, Uhr JW. Circulating tumor cells in patients with breast cancer dormancy. Clin Cancer Res. 2004 Dec 15;10(24):8152-62. doi: 10.1158/1078-0432.CCR-04-1110. PMID 15623589
- [Background] Leone K, Poggiana C, Zamarchi R. The Interplay between Circulating Tumor Cells and the Immune System: From Immune Escape to Cancer Immunotherapy. Diagnostics (Basel). 2018 Aug 30;8(3):59. doi: 10.3390/diagnostics8030059. PMID 30200242
- [Background] Alix-Panabieres C, Pantel K. Liquid Biopsy: From Discovery to Clinical Application. Cancer Discov. 2021 Apr;11(4):858-873. doi: 10.1158/2159-8290.CD-20-1311. PMID 33811121
- [Background] Alix-Panabieres C. The future of liquid biopsy. Nature. 2020 Mar;579(7800):S9. doi: 10.1038/d41586-020-00844-5. No abstract available. PMID 32214259
- [Background] Eslami-S Z, Cortes-Hernandez LE, Alix-Panabieres C. The Metastatic Cascade as the Basis for Liquid Biopsy Development. Front Oncol. 2020 Jul 21;10:1055. doi: 10.3389/fonc.2020.01055. eCollection 2020. PMID 32850309
- [Background] Mego M, Gao H, Cohen EN, Anfossi S, Giordano A, Sanda T, Fouad TM, De Giorgi U, Giuliano M, Woodward WA, Alvarez RH, Valero V, Ueno NT, Hortobagyi GN, Cristofanilli M, Reuben JM. Circulating Tumor Cells (CTC) Are Associated with Defects in Adaptive Immunity in Patients with Inflammatory Breast Cancer. J Cancer. 2016 Jun 3;7(9):1095-104. doi: 10.7150/jca.13098. eCollection 2016. PMID 27326253
- [Background] Ye L, Zhang F, Li H, Yang L, Lv T, Gu W, Song Y. Circulating Tumor Cells Were Associated with the Number of T Lymphocyte Subsets and NK Cells in Peripheral Blood in Advanced Non-Small-Cell Lung Cancer. Dis Markers. 2017;2017:5727815. doi: 10.1155/2017/5727815. Epub 2017 Dec 24. PMID 29434410
- [Background] Mazel M, Jacot W, Pantel K, Bartkowiak K, Topart D, Cayrefourcq L, Rossille D, Maudelonde T, Fest T, Alix-Panabieres C. Frequent expression of PD-L1 on circulating breast cancer cells. Mol Oncol. 2015 Nov;9(9):1773-82. doi: 10.1016/j.molonc.2015.05.009. Epub 2015 Jun 9. PMID 26093818
- [Background] Bergmann S, Coym A, Ott L, Soave A, Rink M, Janning M, Stoupiec M, Coith C, Peine S, von Amsberg G, Pantel K, Riethdorf S. Evaluation of PD-L1 expression on circulating tumor cells (CTCs) in patients with advanced urothelial carcinoma (UC). Oncoimmunology. 2020 Mar 23;9(1):1738798. doi: 10.1080/2162402X.2020.1738798. eCollection 2020. PMID 32391189
- [Background] Darga EP, Dolce EM, Fang F, Kidwell KM, Gersch CL, Kregel S, Thomas DG, Gill A, Brown ME, Gross S, Connelly M, Holinstat M, Cobain EF, Rae JM, Hayes DF, Paoletti C. PD-L1 expression on circulating tumor cells and platelets in patients with metastatic breast cancer. PLoS One. 2021 Nov 15;16(11):e0260124. doi: 10.1371/journal.pone.0260124. eCollection 2021. PMID 34780566
- [Background] Strati A, Koutsodontis G, Papaxoinis G, Angelidis I, Zavridou M, Economopoulou P, Kotsantis I, Avgeris M, Mazel M, Perisanidis C, Sasaki C, Alix-Panabieres C, Lianidou E, Psyrri A. Prognostic significance of PD-L1 expression on circulating tumor cells in patients with head and neck squamous cell carcinoma. Ann Oncol. 2017 Aug 1;28(8):1923-1933. doi: 10.1093/annonc/mdx206. PMID 28838214
- [Background] Jacot W, Mazel M, Mollevi C, Pouderoux S, D'Hondt V, Cayrefourcq L, Bourgier C, Boissiere-Michot F, Berrabah F, Lopez-Crapez E, Bidard FC, Viala M, Maudelonde T, Guiu S, Alix-Panabieres C. Clinical Correlations of Programmed Cell Death Ligand 1 Status in Liquid and Standard Biopsies in Breast Cancer. Clin Chem. 2020 Aug 1;66(8):1093-1101. doi: 10.1093/clinchem/hvaa121. PMID 32712650
- [Background] Sinoquet L, Jacot W, Gauthier L, Pouderoux S, Viala M, Cayrefourcq L, Quantin X, Alix-Panabieres C. Programmed Cell Death Ligand 1-Expressing Circulating Tumor Cells: A New Prognostic Biomarker in Non-Small Cell Lung Cancer. Clin Chem. 2021 Nov 1;67(11):1503-1512. doi: 10.1093/clinchem/hvab131. PMID 34355741
- [Background] European Association For The Study Of The Liver; European Organisation For Research And Treatment Of Cancer. EASL-EORTC clinical practice guidelines: management of hepatocellular carcinoma. J Hepatol. 2012 Apr;56(4):908-43. doi: 10.1016/j.jhep.2011.12.001. No abstract available. PMID 22424438
- [Background] Blanc JF, Debaillon-Vesque A, Roth G, Barbare JC, Baumann AS, Boige V, Boudjema K, Bouattour M, Crehange G, Dauvois B, Decaens T, Dewaele F, Farges O, Guiu B, Hollebecque A, Merle P, Selves J, Aparicio T, Ruiz I, Bouche O; Thesaurus National de Cancerologie Digestive (TNCD); Societe Nationale Francaise de Gastroenterologie (SNFGE); Federation Francophone de Cancerologie Digestive (FFCD); Groupe Cooperateur multidisciplinaire en Oncologie (GERCOR); Federation Nationale des Centres de Lutte Contre le Cancer (UNICANCER); Societe Francaise de Chirurgie Digestive (SFCD); Societe Francaise d'Endoscopie Digestive (SFED); Societe Francaise de Radiotherapie Oncologique (SFRO); Association Francaise pour l'Etude du Foie (AFEF). Hepatocellular carcinoma: French Intergroup Clinical Practice Guidelines for diagnosis, treatment and follow-up (SNFGE, FFCD, GERCOR, UNICANCER, SFCD, SFED, SFRO, AFEF, SIAD, SFR/FRI). Clin Res Hepatol Gastroenterol. 2021 Mar;45(2):101590. doi: 10.1016/j.clinre.2020.101590. Epub 2021 Mar 26. PMID 33780876
- [Background] Hack SP, Spahn J, Chen M, Cheng AL, Kaseb A, Kudo M, Lee HC, Yopp A, Chow P, Qin S. IMbrave 050: a Phase III trial of atezolizumab plus bevacizumab in high-risk hepatocellular carcinoma after curative resection or ablation. Future Oncol. 2020 May;16(15):975-989. doi: 10.2217/fon-2020-0162. Epub 2020 Apr 30. PMID 32352320
- [Background] Yang JC, Hu JJ, Li YX, Luo W, Liu JZ, Ye DW. Clinical Applications of Liquid Biopsy in Hepatocellular Carcinoma. Front Oncol. 2022 Feb 8;12:781820. doi: 10.3389/fonc.2022.781820. eCollection 2022. PMID 35211399
- [Background] Ye Q, Ling S, Zheng S, Xu X. Liquid biopsy in hepatocellular carcinoma: circulating tumor cells and circulating tumor DNA. Mol Cancer. 2019 Jul 3;18(1):114. doi: 10.1186/s12943-019-1043-x. PMID 31269959
- [Background] Winograd P, Hou S, Court CM, Lee YT, Chen PJ, Zhu Y, Sadeghi S, Finn RS, Teng PC, Wang JJ, Zhang Z, Liu H, Busuttil RW, Tomlinson JS, Tseng HR, Agopian VG. Hepatocellular Carcinoma-Circulating Tumor Cells Expressing PD-L1 Are Prognostic and Potentially Associated With Response to Checkpoint Inhibitors. Hepatol Commun. 2020 Aug 4;4(10):1527-1540. doi: 10.1002/hep4.1577. eCollection 2020 Oct. PMID 33024921
- [Background] Seymour L, Bogaerts J, Perrone A, Ford R, Schwartz LH, Mandrekar S, Lin NU, Litiere S, Dancey J, Chen A, Hodi FS, Therasse P, Hoekstra OS, Shankar LK, Wolchok JD, Ballinger M, Caramella C, de Vries EGE; RECIST working group. iRECIST: guidelines for response criteria for use in trials testing immunotherapeutics. Lancet Oncol. 2017 Mar;18(3):e143-e152. doi: 10.1016/S1470-2045(17)30074-8. Epub 2017 Mar 2. PMID 28271869
- [Background] Llovet JM, Bru C, Bruix J. Prognosis of hepatocellular carcinoma: the BCLC staging classification. Semin Liver Dis. 1999;19(3):329-38. doi: 10.1055/s-2007-1007122. PMID 10518312
- [Background] Zhou Y, Wang B, Wu J, Zhang C, Zhou Y, Yang X, Zhou J, Guo W, Fan J. Association of preoperative EpCAM Circulating Tumor Cells and peripheral Treg cell levels with early recurrence of hepatocellular carcinoma following radical hepatic resection. BMC Cancer. 2016 Jul 20;16:506. doi: 10.1186/s12885-016-2526-4. PMID 27439521
- [Background] Su K, Guo L, He K, Rao M, Zhang J, Yang X, Huang W, Gu T, Xu K, Liu Y, Wang J, Chen J, Wu Z, Hu L, Zeng H, Li H, Tong J, Li X, Yang Y, Liu H, Xu Y, Tan Z, Tang X, Feng X, Chen S, Yang B, Jin H, Zhu L, Li B, Han Y. PD-L1 expression on circulating tumor cells can be a predictive biomarker to PD-1 inhibitors combined with radiotherapy and antiangiogenic therapy in advanced hepatocellular carcinoma. Front Oncol. 2022 Aug 2;12:873830. doi: 10.3389/fonc.2022.873830. eCollection 2022. PMID 35982979
- [Background] Chernyak V, Fowler KJ, Kamaya A, Kielar AZ, Elsayes KM, Bashir MR, Kono Y, Do RK, Mitchell DG, Singal AG, Tang A, Sirlin CB. Liver Imaging Reporting and Data System (LI-RADS) Version 2018: Imaging of Hepatocellular Carcinoma in At-Risk Patients. Radiology. 2018 Dec;289(3):816-830. doi: 10.1148/radiol.2018181494. Epub 2018 Sep 25. PMID 30251931